CLINICAL TRIAL: NCT02413060
Title: The Impact of Resistance Training on Type 2 Diabetes Patients.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Yiming Li, Department of endocrinology, Huashan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 42500653-9
Record Dates: First submitted 2015-03-26; First posted 2015-04-09 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Resistance Training

ARMS (2):
- Resistance training (Experimental): Patients of treatment group will undergo resistance training every week sessions
  Interventions: Other: Resistance training; Behavioral: Lifestyle counselling
- Lifestyle counseling (Other): Patients of control group will get the lifestyle counseling every 3 month
  Interventions: Behavioral: Lifestyle counselling

INTERVENTIONS:
Other: Resistance training — This training consists 4 exercises and every exercises lasts 5 seconds.
  Arms: Resistance training
Behavioral: Lifestyle counselling — Lifestyle counselling mainly indicates dietary instruction.

SUMMARY:
The purpose of this study is to determine whether the long-term effects of high-intensity progressive resistance training could improve glucose and lipid metabolism in chinese type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* established type 2 diabetes

Exclusion Criteria:

* severe joint cardiovascular and respiratory system disease, uncontrolled hypertension (160/90 mmHg), severe diabetic nephropathy and neuropathy
* with severe liver and kidney dysfunction
* with mental system disease
* pregnant women or nursing mothers

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-01 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
HbA1c | up to six months

CONTACTS AND LOCATIONS:
Locations (1):
- Cao jia du community health service centre, Shanghai, Shanghai Municipality, China